CLINICAL TRIAL: NCT00170534
Title: An Intervention for Male STD Patients in India
Brief Title: Intervention for Male STDs in India
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 02-106
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2009-04

CONDITIONS: Sexually Transmitted Infection
Keywords: India, male, sexually transmitted infection, STI, STD
MeSH Terms: conditions — Sexually Transmitted Diseases

INTERVENTIONS:
Behavioral: Behavior

SUMMARY:
The specific aim of this study is to complete an ongoing randomized controlled trial of the efficacy of behavioral intervention compared to STI treatment/HIV counseling alone in decreasing risk behavior and incident HIV/STI infections in Mumbai, India.

DETAILED DESCRIPTION:
India has the second highest number of HIV infections of any country in the world, and the epidemic continues unabated. This trial is focused on high risk men attending public STI clinics. A proposed 2 and a half year study, this trial will utilize the continuation of a randomized controlled trial of a behavioral intervention compared to HIV C&T and STI treatment alone targeting HIV uninfected male STI patients. The specific aims are to complete the current behavioral intervention trial and to expand the current investigations to include: the evaluation of men who have sex with men as well as women and evaluate the use of alcohol to the entire sample of recruited men. STI patients will be recruited from three sites and if randomized will agree to a 12 month participation commitment. Strategies employed in both arms of the trial are simple and the fundamental components of an HIV prevention strategy. By demonstrating their effectiveness in India the hope is to encourage the public health leadership to adopt them and continue to change drug treatment availability.

ELIGIBILITY:
Inclusion Criteria:

1. Males, over 16 years of age
2. Hindu or Marathi speakers
3. Have no plan to move permanently out of Mumbia in the following 12 months
4. have a symptom of an STI or have had a sexual exposure in the past 6 months. A sexual exposure is defined as having sex with a commercial sex worker (FSW), having unprotected sex with anyone, male or female, or if the patient came to the clinic seeking an HIV test.
5. Patients will be required to provide an address that can be located by a tracer.

Exclusion Criteria:

1. HIV positive subjects.

Min Age: 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1892
Dates: Start 2004-10; Study Completion 2007-04

CONTACTS AND LOCATIONS:
Locations (1):
- Lokmanya Tilak Municipal General Hospital, Mumbai, India